CLINICAL TRIAL: NCT00345267
Title: Cluster Randomised Controlled Trial of the Effect of the Introduction of an Acute Wheeze/Asthma Integrated Care Pathway on Patient Outcome
Brief Title: Effect of an Integrated Care Pathway on Asthma Care in Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Roche Educational Grant (Unknown); Edinburgh Sick Kids Friends Foundation (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04/S1103/16
Record Dates: First submitted 2006-06-26; First posted 2006-06-28 (Estimated); Last update posted 2006-06-28 (Estimated); Status verified 2006-06

CONDITIONS: Asthma
Keywords: Asthma; Children; Integrated Care Pathway; Evidence based medicine; Prescribing errors
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Device: Integrated Care Pathway

SUMMARY:
Integrated care pathways (ICP) coalesce medical and nursing work practices, unifying and directing care in line with current best practice and guidelines. We wish to examine the introduction of an ICP for children with wheeze/asthma admitted to our hospital. We will determine whether more rigid, but guided care results in faster recovery, quicker discharge with better education and fewer prescribing errors, but also determine whether staff feel alienated by the rigidity of practice, and parents perceive any benefit to the changes introduced.This will be a cluster randomised trial (random weeks) of standard or ICP care in 180 patients admitted to Sick Kids with wheeze/asthma. Parents will be asked to complete a questionnaire on admission and contacted at 10-14 days post discharge and asked to recall education provided at discharge; no other patient or parent intervention will be required.It is expected to take 40 weeks to recruit 180 patients.

DETAILED DESCRIPTION:
Children admitted to hospital with wheeze/asthma are provided with care by a large number of clinicians with varying levels of skills and experiences. Providing a uniform, safe level of care, according to evidence based guidelines is challenging given the levels of experience within each hospital. Integrated care pathways are a multidisciplinary document incorporating medical, nursing, pharmacy and observational charts within a single chronological document. The study is to assess whether such documents can speed recovery and discharge, with care adhering more closely to evidence based guidelines for treatment and education. In addition we wish to assess patient safety (through prescribing errors) and parental and staff attitudes to the ICP introduction. Children arriving at the emergency department will be provided with care by either intergrated care pathway or standard care in 7 day clusters, randomised in 8 week blocks.

Comparison: We will compare the time from arrival at hospital to discharge from the ward as our primary outcome.

Other comparisons to be made for: Speed of recovery of heart rate and respiratory rate Time to require no supplemental oxygen Time to achieve 4 hourly spacing of bronchodilator Number and degree of prescribing errors Provision of education to parents Provision of care adhering to asthma guidelines (accurate discharge dose of prednisolone from emergency dept, use of multidose salbutamol rather than nebuliser) Number of clinical contacts required with patients Staff opinion of ICP before and after introduction Parental opinion of care in different groups Parental recall of advice/education provided to them during admission Possible Hawthorne effect during period of the study

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-16 years (inclusive) arriving at the Emergency Department with acute wheeze/asthma

Exclusion Criteria:

* Children requiring high dependency care
* Children with significant neurological or cardiac disease

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180
Dates: Start 2004-08; Study Completion 2005-03

PRIMARY OUTCOMES:
Length of stay in hospital

SECONDARY OUTCOMES:
Speed of recovery of heart rate and respiratory rate
Time to require no supplemental oxygen
Time to achieve 4 hourly spacing of bronchodilator
Number and degree of prescribing errors
Provision of education to parents
Provision of care adhering to asthma guidelines (accurate discharge dose of prednisolone from emergency dept, use of multidose salbutamol rather than nebuliser)
Number of clinical contacts required with patients
Staff opinion of ICP before and after introduction
Parental opinion of care in different groups
Parental recall of advice/education provided to them during admission
Possible Hawthorne effect during period of the study
Parental recall of advice to contact primary care

CONTACTS AND LOCATIONS:
Overall Officials: Steve Cunningham, MD, PhD, Study Director — University of Edinburgh; Robin Prescott, PhD, FRCP, Study Director — University of Edinburgh
Locations (1):
- Dept of Respiratory and Sleep Medicine, Royal Hospital for Sick Children, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Derived] Cunningham S, Logan C, Lockerbie L, Dunn MJ, McMurray A, Prescott RJ. Effect of an integrated care pathway on acute asthma/wheeze in children attending hospital: cluster randomized trial. J Pediatr. 2008 Mar;152(3):315-20. doi: 10.1016/j.jpeds.2007.09.033. Epub 2007 Nov 26. PMID 18280833